CLINICAL TRIAL: NCT01917734
Title: Evaluation of the Effectiveness of an Integrated Program for the Management of Severe Acute Malnutrition in Children in Madhya Pradesh, India
Brief Title: Integrated Program for Children With Severe Acute Malnutrition in Madhya Pradesh, India
Status: Completed | Type: Observational
Sponsor: Victor M. Aguayo (Other)
Collaborators: Gandhi Medical College, Bhopal (Other); Bundelkhand Medical College, Sagar, Madhya Pradesh (Unknown); Gajara Raja Medical College (Other)
Responsible Party: Sponsor-Investigator, Victor M. Aguayo, Chief, Child Nutrition and Development, India, UNICEF
Organization: UNICEF (Other)
Other Study IDs: MP-SAM-2010
Record Dates: First submitted 2013-08-03; First posted 2013-08-07 (Estimated); Last update posted 2013-08-07 (Estimated); Status verified 2013-08

CONDITIONS: Severe Malnutrition
Keywords: severe acute malnutrition; severe wasting; facility-based care; community-based care; Madhya Pradesh; India
MeSH Terms: conditions — Malnutrition; Severe Acute Malnutrition; Cachexia | interventions — S-Adenosylmethionine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- IM-SAM: Children 6-59 months with bilateral pitting edema, and/or WHZ < - 3 and/or MUAC < 115 mm.
  Interventions: Other: Therapeutic feeding for children with SAM

INTERVENTIONS:
Other: Therapeutic feeding for children with SAM — Comparison of outcomes between children with complicated SAM and children with uncomplicated SAM as well as comparisn of outcomes against national and internationally agreed upon standards of care

SUMMARY:
The purpose of this study is to assesses the effectiveness of an integrated model for the management of severe acute malnutrition (IM-SAM) in India comprising facility- and community-based care and using locally-adapted protocols

DETAILED DESCRIPTION:
Madhya Pradesh's program for the provision of care to children with severe acute malnutrition (SAM) was initiated in the district of Shivpuri in January 2006. By January 1, 2010, Madhya Pradesh National Rural Health Mission (NRHM) had established 199 Nutrition Rehabilitation Centers (NRCs) where children were receiving therapeutic care following protocols based on the guidelines for the management of SAM by the World Health Organization (WHO)and the Indian Academy of Pediatrics.

The detection of children with SAM was ensured in the communities by frontline workers in the context of monthly growth monitoring and promotion sessions. Once at the NRC the age, weight, height, mid-upper arm circumference (MUAC) and presence of bilateral pitting edema were determined for each child. SAM was defined as per WHO recommendations by the presence of bilateral pitting edema or the presence of severe wasting. Severe wasting was defined by a MUAC below 115 mm and/or a weight-for-height z-score (WHZ) < - 3 of the median WHZ in WHO Child Growth Standards. All children 6-59 months with bilateral pitting edema, and/or WHZ < - 3 and/or MUAC < 115 mm were admitted to the NRC.

Once children were admitted to the NRC, a medical doctor conducted a clinical examination on them to detect the presence of medical complications (lethargy, pneumonia, dehydration, fever, tuberculosis, and/or severe anemia) using the criteria for the Integrated Management of Neonatal and Childhood Illnesses (IMNCI).

As per protocol, children with edema, and/or medical complications, and/or poor appetite were fed locally-prepared F-75 therapeutic milk every two hours for 48 hours (stabilization phase) while their medical complications were treated. After completion of the initial 48 hours, children were fed alternatively F-75 and locally-prepared F-100 therapeutic milk six times a day for about 48 hours (transition phase). After the transition phase, children were fed F-100 and locally-produced lipid-based therapeutic food (TF) with the aims of initiating rapid weight gain (rehabilitation phase). Children with normal appetite and free of medical complications entered the rehabilitation phase from the day of admission. All children received a course of broad spectrum antibiotic.

Upon the completion of a prescribed 14-day stay in the NRC, children were transitioned to the community phase of the program where they were followed up by community-based frontline workers. Frontline workers were to ensure that the child benefited a Supplementary Nutrition Program (SNP) and returned for a follow up visit at the NRC every 15 days during the 60 days following discharge. At the four follow up visits, children's weight gain was assessed and mothers were counseled on child feeding and care.

From January 1 to December 31, 2010 a total of 44,017 children 6-59 months old were admitted to the IM-SAM program. This study evaluates the effectiveness of the program by analyzing program outcomes in sample of children (n=2,740) randomly selected among the 44,017 children admitted.

ELIGIBILITY:
Inclusion Criteria:

* Age 6-59 months
* Clinical diagnosis of with bilateral pitting oedema
* Anthropometric diagnosis of severe wasting (WHZ < - 3 and/or MUAC < 115 mm)

Exclusion Criteria:

* Severe congenital conditions whose clinical management required highly specialized skills only available ar the district hospital
* Severe pathological conditions whose clinical management required highly specialized skills only available ar the district hospital

Ages: 6 Months to 59 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: The detection of children with severe acute malnutrition was ensured in the communities by frontline workers in the context of monthly growth monitoring and promotion sessions.
Sampling Method: Probability Sample
Enrollment: 2740 (Actual)
Dates: Start 2010-01; Primary Completion 2011-12 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Recovery | 74 days
  Weight gain >= 15% of initial weight gain
Discharged | 74 days
  Proportion of children completing a 14-day stay in the NRC, transitioned to the community phase of the program and atteding at least two of the four community-based follow up visits.

SECONDARY OUTCOMES:
Weight gain | 74 days
  Average weight gain per Kg body mass per day during stay in the programme

OTHER OUTCOMES:
Discharged | 74 days
  Completed treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Atal Bal State Nutrition Mission and National Rural Health Mission, Bhopal, Madhya Pradesh, India

REFERENCES:
- [Derived] Aguayo VM, Agarwal V, Agnani M, Das Agrawal D, Bhambhal S, Rawat AK, Gaur A, Garg A, Badgaiyan N, Singh K. Integrated program achieves good survival but moderate recovery rates among children with severe acute malnutrition in India. Am J Clin Nutr. 2013 Nov;98(5):1335-42. doi: 10.3945/ajcn.112.054080. Epub 2013 Sep 25. PMID 24067666